CLINICAL TRIAL: NCT05219500
Title: PSMA-directed Targeted Alpha Therapy With FPI-2265 (225Ac-PSMA-I&T) for the Treatment of Metastatic Castration-resISTant Prostate Cancer (TATCIST). A Phase II Clinical Trial.
Brief Title: Targeted Alpha Therapy With 225Actinium-Prostate Specific Membrane Antigen (PSMA)-I&T of Castration-resISTant Prostate Cancer (TATCIST).
Acronym: TATCIST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fusion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPI-2265-201
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FPI-2265 (Experimental): All patients will receive FPI-2265, administered at 8 ± 1-week interval, with the initial activity of 100 kBq/kg (±10%).
  Interventions: Drug: FPI-2265

INTERVENTIONS:
Drug: FPI-2265 — Small molecule capable of binding to the domain of PSMA radiolabeled with Ac225
  Other Names: Ac225-PSMA I&T

SUMMARY:
The treatment regimen will consist of 4 doses of FPI-2265

DETAILED DESCRIPTION:
The treatment regimen will consist of 4 doses of FPI-2265, administered at 8 ± 1 week intervals, with an initial activity of 100 kilobecquerel (kBq)/kg (±10%).

Additional doses will be administered at 100 kBq/kg (±10%) with the following exceptions:

* Participants who experience dose-modifying events.
* Participants with a confirmed decline in PSA>=50%.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥ 18 years.
2. Participants must have the ability to understand and sign an approved informed consent (ICF).
3. Participants must have the ability to understand and comply with all protocol requirements.
4. Adenocarcinoma of prostate proven by histopathology.
5. Life expectancy of 6 months or more.
6. Unresectable metastases.
7. Documented progressive disease (PD); progressive mCRPC will be based on at least 1 of the following criteria:

   1. Serum PSA progression is defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal starting value is 1.0 ng/mL, if PSA is the only indication of progression.
   2. Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions.
   3. Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan (2+2 PCWG3 criteria).
8. If known Breast Cancer gene (BRCA) mutations are present, participants should have received FDA approved therapies such as poly-ADP ribose polymerase (PARP) inhibitors and progressed.
9. Castration resistant disease with confirmed testosterone level ≤ 50 ng/dL under prior androgen deprivation therapy (ADT). Must have a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L).
10. Positive PSMA PET/CT scans, obtained with approved PSMA-ligands, defined as at least one PSMA-positive metastatic lesion and no PSMA-negative lesions.
11. ECOG-PS 0 to 1.
12. Hemoglobin (Hgb) concentration ≥ 9.0 g/dL.
13. Platelet counts ≥ 100 × 10^9/L.
14. White blood cell (WBC) count ≥ 2.0 × 10^9/L, absolute neutrophil count (ANC) > 1.5 × 10^9/L.

    a. Hematological criteria cannot be met with ongoing or recent blood transfusions (within 7 days prior to the scheduled first dose of study treatment) or require growth factor support (within 21 days prior to the scheduled first dose of study treatment).
15. Alanine aminotransferase or aspartate aminotransferase ≤ 3.0 × upper limit of normal (ULN).
16. Serum total bilirubin ≤ 1.5 × ULN; in participants with Gilbert's syndrome, a total bilirubin ≤ 3 times ULN and direct bilirubin within normal limits are permitted.
17. Albumin ≥ 2.5 g/dL.
18. Serum/plasma creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min based on the Cockcroft-Gault formula.
19. Prothrombin time, international normalized ratio or prothrombin time test < 1.5 × ULN.
20. Received ≥ 1 androgen receptor axis-targeted therapies (ARAT).
21. Participants on anti-androgen therapy are allowed to continue their treatment at the discretion of their treating physician.

Exclusion Criteria:

1. Less than 6 weeks from enrollment since last myelosuppressive therapy (including Docetaxel, Cabazitaxel, 223Ra, 153Sm, 177Lu-PSMA-617/other Lu-PSMA RLT or any other radionuclide therapy). Participants who received previous treatment with Ac-225 are excluded.
2. Participants who received more than 4 prior lines of systemic therapy for CRPC.
3. Urinary tract obstruction as evidenced by Tc-99m DTPA renal scan with diuretics.
4. Participants with skeletal metastases presenting as a superscan on a 99m Tc MDP Bone Scan.

   Superscan is defined as a bone scan which demonstrates markedly increased skeletal radioisotope uptake relative to soft tissues in association with absent or faint renal activity (absent kidney sign).
5. Persistent baseline dry eye or dry mouth > Grade 1 from prior RLT.
6. Persistent prior AEs > Grade 1 from prior anti-cancer therapies.
7. Abnormal renal function (estimated glomerular filtration rate < 60 mL/min), baseline Hgb < 9g/dL, ANC < 1.5 ×10^9/L, platelets < 100 ×10^9/L, and prothrombin time, international normalized ratio or prothrombin time test ≥ 1.5 × ULN.
8. Administration of an investigational agent ≤ 60 days or 5 half-lives, whichever is shorter, prior to Cycle 1, Week 0.
9. Known presence of central nervous system (CNS) metastases or liver metastases.
10. Active malignancy other than low-grade non-muscle-invasive bladder cancer and non-melanoma skin cancer.
11. Concurrent illness that may jeopardize the participant's ability to undergo study procedures as determined by the Investigator.
12. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
13. Concurrent serious (as determined by the investigator) medical conditions, including, but not limited to, New York Heart Association Class III or IV congestive heart failure, unstable ischemia, uncontrolled symptomatic arrhythmia, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
14. Major surgery ≤ 30 days prior to enrollment.
15. Planning to conceive pregnancy during the treatment and up to 6 months after the last treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of FPI-2265 on prostate-specific antigen (PSA) in participants with mCRPC. | From start of treatment until 12 weeks after the first treatment.
  Frequency and proportion of participants with PSA50, defined as ≥ 50% decline in PSA level by 12-weeks after the first treatment.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of FPI- 2265. | From first treatment dose to up to 24 months after last treatment.
  * Frequency, duration and severity of treatment emergent adverse events (TEAEs) evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0).
  * Changes in clinical laboratory, electrocardiograms (ECGs) and physical examinations compared to baseline.
To evaluate the anti-tumor activity of FPI-2265. | From first treatment until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 24 months after last treatment.
  * Maximum % PSA decline.
  * PSA progression free survival (PFS).
  * Time to best PSA response
  * Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
  * Disease control rate (DCR) per RECIST v1.1.
  * Duration of response (DoR) based on RECIST v1.1/Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.
  * Radiographic progression-free survival (rPFS) per PCWG3 criteria.
  * Overall survival (OS).
To assess the impact of FPI-2265 on participant reported outcomes. | From first treatment until 24 months after last treatment.
  * The frequency and proportion of participants with an improvement in bone pain levels.
  * Change in quality of life (QoL) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Barnett, Study Director — Fusion Pharmaceuticals Inc.
Locations (2):
- United States (2):
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas